CLINICAL TRIAL: NCT06190314
Title: SERUM VITAMIN B12 LEVELS IN PATIENTS WITH HEMORRHAGIC VS ISCHEMIC CEREBROVASCULAR EVENT.
Acronym: ViBEVC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital General de Mexicali (Other)
Collaborators: Sandoval Briones Jocelin Lisset (Unknown); Hirata Medina Nancy Midory (Unknown); Felix Escobedo Marisol (Unknown); Cervantes De Carlos Cereza Guadalpe (Unknown); Aceves Lozano Natalia (Unknown); Cota Andara Manuel Eduardo (Unknown); Avila Pacheco Manlio Abraham (Unknown); Rodriguez Gonzalez Alondra (Unknown); Barruquin Sandoval Claudia Pamela (Unknown); González Gómez René Ignacio (Unknown); Jaramillo Ramirez Hiram Javier. (Unknown)
Responsible Party: Principal Investigator, Hiram Jaramillo Ramirez, Serum Vitamin B12 levels in patients with hemorrhagic vs ischemic cerebrovascular event, Hospital General de Mexicali
Other Study IDs: 02-01-HGMXL/CEI/2023-23
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Cerebrovascular Event; Vitamin b12; Hemorrhagic Stroke; Ischemic Stroke
Keywords: Stroke; Hemorrhagic; B12; Ischemic
MeSH Terms: conditions — Hemorrhagic Stroke; Ischemic Stroke; Stroke; Ischemia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — blood serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with ischemic stroke: measure serum vitamin b12 levels
  Interventions: Diagnostic Test: Measure serum vitamin b12 levels
- patients with hemorrhagic stroke: measure serum vitamin b12 levels
  Interventions: Diagnostic Test: Measure serum vitamin b12 levels

INTERVENTIONS:
Diagnostic Test: Measure serum vitamin b12 levels — Measure the vitamin b-12 levels in patients that are admitted for stroke of any kind

SUMMARY:
Cerebral vascular events (CVA) have a high prevalence in our environment; they are the first cause of disability and the second cause of death in the world (6.6 million deaths). 71% of all strokes worldwide correspond to the ischemic type, which is defined as an infarction in the brain, spinal cord or retina; The remaining 10-40% are hemorrhagic and are due to rupture of cerebral arteries. Until epidemiological week 35 of 2022, 34,643 cases were reported in Mexico, for this week in 2021, 26,462 cases had been reported. Baja California is among the first three places in the country with the highest number of reported cases, the majority corresponding to the male sex. The key clinical characteristic is the sudden appearance of a focal neurological deficit. Imaging studies such as head computed tomography or magnetic resonance imaging allow us to differentiate the subtype and mechanism of CVD since treatment differs markedly between CVD of ischemic origin and that of hemorrhagic origin. Vitamin B12 or cobalamin is a tetrapyrrole cofactor; One of its functions is to participate in the metabolism of homocysteine, which has been reported in various studies and it has been shown that high levels of this increase the risk of vascular diseases, such as stroke. On the other hand, vitamin B12 deficiency can lead to platelet dysfunction, causing significant bleeding. There are few protocols that have sought the direct association of cobalamin with CVD and even fewer with the hemorrhagic type. This condition is one of the main causes of admission to the Emergency Service of the General Hospital of Mexicali where they are given the necessary attention such as performing imaging studies and taking laboratory samples and based on the results the treatment to be followed is decided; However, measurements of vitamin B12 levels are not performed in this population. If the association is demonstrated, it could be implemented as a preventive measure for cerebral vascular events.

DETAILED DESCRIPTION:
General objective: To demonstrate if there is a difference between serum levels of vitamin B12 in patients with hemorrhagic cerebral vascular event compared to patients with ischemic cerebral vascular event.

Specific objectives

* Describe the characteristics of the study population (sex, age, comorbidities, laboratory diagnoses)
* Determine serum levels of vitamin B12 in patients with cerebral vascular event
* Establish the prevalence of vitamin B12 deficiency in patients with cerebral vascular events.
* Correlations of vitamin B12 deficiency with the severity of the disease
* To establish whether there is a difference in serum vitamin B12 levels between patients with ischemic stroke compared to hemorrhagic stroke.
* Determine if the degree of deficiency correlates with mortality
* Compare vitamin B12 levels by subgroups

STUDY DESIGN This will be a prospective, observational, analytical study of patients admitted to the General Hospital of Mexicali with a diagnosis of ischemic or hemorrhagic stroke.

SOURCE FOR OBTAINING PATIENTS Patients admitted to the adult emergency department of the Mexicali General Hospital with a diagnosis of ischemic or hemorrhagic stroke are included. The information will be collected from the electronic clinical record.

Non-probability sampling for convenience. Select all patients who arrive at the hospital who meet inclusion criteria and do not have any exclusion or elimination criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Have a diagnosis of a cerebral vascular event
* Being a hospitalized patient at the General Hospital of Mexicali

Exclusion Criteria:

* Patients without lab tests during their hospitalization
* Patients without a cranial CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Select all patients who arrive at the hospital who meet inclusion criteria and do not have any exclusion or elimination criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Difference of vitamin B12 level between ischemic and hemorrhagic stroke | November 2023 - November 2024
  Demonstrate if there is a difference between serum levels of vitamin B12 in patients with hemorrhagic cerebral vascular event compared to patients with ischemic cerebral vascular event.

SECONDARY OUTCOMES:
Vitamin B12 defficiency in patients with stroke | November 2023 - November 2024
  Vitamin B12 defficiency in patients with any kind of stroke
Population characteristics | November 2023 - November 2024
  Determine if variables like sex, age, comorbilities and lab tests have a correlation between stroke and Vitamin B12 levels
Mortality and vitamin B 12 deficiency in this specific population | November 2023 - November 2024
  Analize the levels of vitamin B12 and the in-hospital mortality in this population
Levels of B12 vitamin and severity of stroke | November 2023 - November 2024
  Analize if there is a significant difference between the levels of B12 and the severity of stroke

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Mexicali, Mexicali, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed S, Bogiatzi C, Hackam DG, Rutledge AC, Sposato LA, Khaw A, Mandzia J, Azarpazhoo MR, Hachinski V, Spence JD. Vitamin B 12 deficiency and hyperhomocysteinaemia in outpatients with stroke or transient ischaemic attack: a cohort study at an academic medical centre. BMJ Open. 2019 Jan 21;9(1):e026564. doi: 10.1136/bmjopen-2018-026564. PMID 30670531
- [Background] Arch AE, Weisman DC, Coca S, Nystrom KV, Wira CR 3rd, Schindler JL. Missed Ischemic Stroke Diagnosis in the Emergency Department by Emergency Medicine and Neurology Services. Stroke. 2016 Mar;47(3):668-73. doi: 10.1161/STROKEAHA.115.010613. Epub 2016 Feb 4. PMID 26846858
- [Background] Bick RL. Platelet function defects associated with hemorrhage or thrombosis. Med Clin North Am. 1994 May;78(3):577-607. doi: 10.1016/s0025-7125(16)30148-1. PMID 8170260
- [Background] Bjorklund G, Peana M, Dadar M, Lozynska I, Chirumbolo S, Lysiuk R, Lenchyk L, Upyr T, Severin B. The role of B vitamins in stroke prevention. Crit Rev Food Sci Nutr. 2022;62(20):5462-5475. doi: 10.1080/10408398.2021.1885341. Epub 2021 Mar 16. PMID 33724098
- [Background] Campbell BCV, De Silva DA, Macleod MR, Coutts SB, Schwamm LH, Davis SM, Donnan GA. Ischaemic stroke. Nat Rev Dis Primers. 2019 Oct 10;5(1):70. doi: 10.1038/s41572-019-0118-8. PMID 31601801
- [Background] Campbell BCV, Khatri P. Stroke. Lancet. 2020 Jul 11;396(10244):129-142. doi: 10.1016/S0140-6736(20)31179-X. PMID 32653056
- [Background] Castro R, Rivera I, Blom HJ, Jakobs C, Tavares de Almeida I. Homocysteine metabolism, hyperhomocysteinaemia and vascular disease: an overview. J Inherit Metab Dis. 2006 Feb;29(1):3-20. doi: 10.1007/s10545-006-0106-5. PMID 16601863
- [Background] Chatthanawaree W. Biomarkers of cobalamin (vitamin B12) deficiency and its application. J Nutr Health Aging. 2011 Mar;15(3):227-31. doi: 10.1007/s12603-010-0280-x. PMID 21369672
- [Background] Clarke R, Halsey J, Lewington S, Lonn E, Armitage J, Manson JE, Bonaa KH, Spence JD, Nygard O, Jamison R, Gaziano JM, Guarino P, Bennett D, Mir F, Peto R, Collins R; B-Vitamin Treatment Trialists' Collaboration. Effects of lowering homocysteine levels with B vitamins on cardiovascular disease, cancer, and cause-specific mortality: Meta-analysis of 8 randomized trials involving 37 485 individuals. Arch Intern Med. 2010 Oct 11;170(18):1622-31. doi: 10.1001/archinternmed.2010.348. PMID 20937919
- [Background] Devalia V, Hamilton MS, Molloy AM; British Committee for Standards in Haematology. Guidelines for the diagnosis and treatment of cobalamin and folate disorders. Br J Haematol. 2014 Aug;166(4):496-513. doi: 10.1111/bjh.12959. Epub 2014 Jun 18. PMID 24942828
- [Background] Dong H, Pi F, Ding Z, Chen W, Pang S, Dong W, Zhang Q. Efficacy of Supplementation with B Vitamins for Stroke Prevention: A Network Meta-Analysis of Randomized Controlled Trials. PLoS One. 2015 Sep 10;10(9):e0137533. doi: 10.1371/journal.pone.0137533. eCollection 2015. PMID 26355679
- [Background] Dudi, Parmila, Anita Rani, Bela Goyal, Geeta Kampani, Kamlesh Rabari, Ashish Kothari, and Sarama Saha. "Association of Vitamin B12 Transporter Protein (Transcobalamin II) Genetic Polymorphisms with Risk of Stroke: An Observational Pilot Study in North Indian Population." Meta Gene 25 (September 2020): 100747. https://doi.org/10.1016/j.mgene.2020.100747.
- [Background] Duschek N, Basic J, Falkensammer J, Taher F, Assadian A. B-Vitamin Serum Concentrations Predicting Long-Term Overall and Stroke-Free Survival after Carotid Endarterectomy. J Stroke Cerebrovasc Dis. 2016 May;25(5):1235-1243. doi: 10.1016/j.jstrokecerebrovasdis.2016.01.044. Epub 2016 Feb 28. PMID 26935113
- [Background] George PM, Steinberg GK. Novel Stroke Therapeutics: Unraveling Stroke Pathophysiology and Its Impact on Clinical Treatments. Neuron. 2015 Jul 15;87(2):297-309. doi: 10.1016/j.neuron.2015.05.041. PMID 26182415
- [Background] Graham IM, Daly LE, Refsum HM, Robinson K, Brattstrom LE, Ueland PM, Palma-Reis RJ, Boers GH, Sheahan RG, Israelsson B, Uiterwaal CS, Meleady R, McMaster D, Verhoef P, Witteman J, Rubba P, Bellet H, Wautrecht JC, de Valk HW, Sales Luis AC, Parrot-Rouland FM, Tan KS, Higgins I, Garcon D, Andria G, et al. Plasma homocysteine as a risk factor for vascular disease. The European Concerted Action Project. JAMA. 1997 Jun 11;277(22):1775-81. doi: 10.1001/jama.1997.03540460039030. PMID 9178790
- [Background] Green R, Allen LH, Bjorke-Monsen AL, Brito A, Gueant JL, Miller JW, Molloy AM, Nexo E, Stabler S, Toh BH, Ueland PM, Yajnik C. Vitamin B12 deficiency. Nat Rev Dis Primers. 2017 Jun 29;3:17040. doi: 10.1038/nrdp.2017.40. PMID 28660890
- [Background] Hand PJ, Kwan J, Lindley RI, Dennis MS, Wardlaw JM. Distinguishing between stroke and mimic at the bedside: the brain attack study. Stroke. 2006 Mar;37(3):769-75. doi: 10.1161/01.STR.0000204041.13466.4c. Epub 2006 Feb 16. PMID 16484610
- [Background] Huang X, Li Y, Li P, Li J, Bao H, Zhang Y, Wang B, Sun N, Wang J, He M, Yin D, Tang G, Chen Y, Cui Y, Huang Y, Hou FF, Qin X, Huo Y, Cheng X. Association between percent decline in serum total homocysteine and risk of first stroke. Neurology. 2017 Nov 14;89(20):2101-2107. doi: 10.1212/WNL.0000000000004648. Epub 2017 Oct 13. PMID 29030456
- See also: Vitamin B 12 deficiency and hyperhomocysteinaemia in outpatients with stroke or transient ischaemic attack: a cohort study at an academic medical centre — https://pubmed.ncbi.nlm.nih.gov/30670531/
- See also: Missed Ischemic Stroke Diagnosis in the Emergency Department by Emergency Medicine and Neurology Services — https://pubmed.ncbi.nlm.nih.gov/26846858/
- See also: Ischaemic stroke — https://www.nature.com/articles/s41572-019-0118-8
- See also: Stroke — https://pubmed.ncbi.nlm.nih.gov/32653056/
- See also: Homocysteine metabolism, hyperhomocysteinaemia and vascular disease: an overview — https://pubmed.ncbi.nlm.nih.gov/16601863/
- See also: Biomarkers of cobalamin (vitamin B12) deficiency and its application — https://link.springer.com/article/10.1007/s12603-010-0280-x
- See also: Guidelines for the diagnosis and treatment of cobalamin and folate disorders — https://pubmed.ncbi.nlm.nih.gov/24942828/
- See also: Efficacy of Supplementation with B Vitamins for Stroke Prevention: A Network Meta-Analysis of Randomized Controlled Trials — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4565665/
- See also: Novel Stroke Therapeutics: Unraveling Stroke Pathophysiology and Its Impact on Clinical Treatments — https://pubmed.ncbi.nlm.nih.gov/26182415/
- See also: Plasma homocysteine as a risk factor for vascular disease. The European Concerted Action Project — https://pubmed.ncbi.nlm.nih.gov/9178790/
- See also: Vitamin B12 deficiency — https://www.nature.com/articles/nrdp201740
- See also: Distinguishing between stroke and mimic at the bedside: the brain attack study — https://pubmed.ncbi.nlm.nih.gov/16484610/
- See also: Efficacy of folic acid therapy in primary prevention of stroke among adults with hypertension in China: the CSPPT randomized clinical trial — https://pubmed.ncbi.nlm.nih.gov/25771069/